CLINICAL TRIAL: NCT06065462
Title: Safety and Efficacy of Targeting PP2A in Ovarian Clear Cell Carcinoma Using Dostarlimab and LB-100
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GSK Pharma (Unknown); Lixte (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1047; NCI-2023-07922 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Clear Cell Carcinoma
MeSH Terms: interventions — dostarlimab; LB100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dostarlimab + LB-100 (Experimental): Dostarlimab will be given by vein over about 30 minutes on Day 1 of each cycle. LB-100 will be given by vein on Days 1-3 of each cycle. The first doses will be given over about 2 hours. After that, doses may be given over as little as 30 minutes.
  Interventions: Drug: Dostarlimab; Drug: LB-100

INTERVENTIONS:
Drug: Dostarlimab — Given by vein (IV)
Drug: LB-100 — GIven by vein (IV)

SUMMARY:
To learn if the combination of dostarlimab and LB-100 can help to control ovarian clear cell carcinoma

DETAILED DESCRIPTION:
Primary Objectives:

1. To estimate overall survival in patients with recurrent ovarian clear cell carcinoma being treated with LB-100 and dostarlimab, including specific survival probabilities at 6 and 12 months.

Secondary Objectives:

1. To describe clinically significant and immune related adverse events (ir-AEs) in the study population.
2. To determine the objective response rate (ORR), time to initial response, progression free survival (PFS), and duration of response (DOR) using modified RECIST v1.1 criteria.

   a. Although the clinical benefit of these drugs has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.
3. Translational:

   1. To describe PP2A activity and immune changes, using baseline and on-treatment tumor biopsies and peripheral blood mononuclear cells (PBMCs)
   2. To describe expression of mismatch repair proteins using immunohistochemistry (IHC)
   3. To correlate circulating tumor DNA (ctDNA) levels with response by modified RECIST v1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be assessed within 28 days of starting study treatment:

1. Ability to provide signed informed consent
2. Age 18-75 years at time of study entry
3. Willingness and ability to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
4. Histology showing recurrent clear cell ovarian, peritoneal, or fallopian tube cancer (mixed histology with predominant clear cell component is acceptable).
5. Receipt of at least one prior line of therapy for recurrent disease or development of platinum resistant or refractory disease, defined by progression of disease on a platinum-containing regimen or recurrence of disease within 180 days of previous platinum treatment
6. Available somatic mutation testing results (CLIA source) that reveal no PPP2R1A mutations
7. Measurable disease based on modified RECIST v1.1. For the purposes of this study measurable disease is defined at least one "target lesion" that can be accurately measured in at least one dimension (longest dimension to be recorded). Each target lesion must be >20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >10 mm when measured by spiral CT. The target lesion must be distinct from other tumor areas selected for pre-treatment biopsies. Second lesion selected for pre-treatment biopsy must be biopsy accessible.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. See Section 14.
9. Life expectantly of ≥12 weeks
10. Adequate normal organ and bone marrow function as defined below.

    1. Hemoglobin ≥8.0 g/ dL
    2. Absolute neutrophil count (ANC) ≥ 1000/mm3
    3. Platelet count ≥100 x 109/L (>100,000/mm3)
    4. Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    5. AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5 x ULN
    6. Measured creatinine clearance (CL) ≥ 50 mL/min or Calculated creatinine CL ≥ 50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
11. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. The effects of dostarlimab and LB-100 on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (See Section 5.6.2).
12. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy)

Exclusion Criteria:

Exclusion criteria will be assessed within 28 days of starting study treatment:

1. Participation in another clinical study with an investigational product (IP) during the last 28 days.
2. Prior treatment with anti-CTLA-4 or anti-PDL-1/PD-1 antibodies.
3. Patients with mismatch repair deficient (dMMR) by IHC or microsatellite instability-high tumors
4. Concurrent treatment on another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
5. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤21 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of the agent, a longer wash-out period will be required, as agreed by study sponsors and the investigators.
6. Any unresolved toxicity NCI CTCAE Grade 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   1. Subjects with Grade 2 neuropathy will be evaluated on a case-by-case basis after consultation with the principal investigator.
   2. Subjects with irreversible toxicity not reasonably expected to be exacerbated by the treatment with investigational therapy may be included only after consultation with the primary investigator.
7. Any concurrent chemotherapy, immunotherapy, or hormonal therapy for cancer treatment.
8. Major surgical procedure (defined by the investigator) within 28 days prior to the first dose of treatment. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic or hematologic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders, including inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis in the last 6 months (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome.

    a. The following exceptions to this criterion are listed below. i. Subjects with vitiligo or alopecia. ii. Subjects with hypothyroidism stable on hormone replacement. iii. Any chronic skin condition that does not require systemic therapy. iv. Subjects without active disease in the last 5 years may be included but only after consultation with the primary investigator.

    v. Subjects with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to: ongoing or active infection; symptomatic congestive heart failure; uncontrolled hypertension; unstable angina pectoris; cardiac arrythmia; interstitial lung disease; chronic obstructive pulmonary disease requiring systemic steroid therapy, oxygen, or hospitalization; serious chronic gastrointestinal conditions associated with diarrhea; or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
12. Any medical, social, or psychological condition that would interfere with evaluation of study treatment or interpretation of participant safety or study results.
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen, or HBsAg, result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).

    1. Subjects with a past or resolved HBV infection (defined as presence of hepatitis B core antibody, or anti-HBc, and absence of HBsAg) are eligible.
    2. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
    3. Patients with positive results of HIV that meet all of the following eligibility criteria may be enrolled:

    i. Have a T-cell (CD4+) count ≥350 cells/µL ii. No history of opportunistic infections or other malignancies iii. Have an HIV viral load less than 400 copies/mL prior to enrollment iv. In the opinion of the investigator, their antiretroviral therapy (ART) or other HIV treatments will not interfere with the activity of the investigational product or cause any confusion with the assessment of the investigational drug toxicities
14. History of another primary malignancy except for the following histories:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of treatment and of low potential risk of recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
15. History of leptomeningeal carcinomatosis.
16. Untreated brain metastases or spinal cord compression. Subjects with suspected brain metastases at screening should have an MRI (preferred) or CT preferably with IV contrast of the brain prior to study entry.

    a. Subjects with treated brain metastasis as evidenced by stable findings on brain MRI performed 4-6 weeks after completion of treatment would be eligible.
17. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of trial therapies. Listed below are the exceptions to this criterion.

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular infection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
19. Receipt of live attenuated vaccine within 30 days prior to the first dose of treatment. Note: subjects, if enrolled, should not receive live vaccines whilst receiving treatment and up to 90 days after the last dose of treatment
20. Female subjects who are pregnant or breastfeeding or of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of treatment

    a. Pregnant women are excluded from this study because the investigational agents have unknown teratogenic or abortifacient effects. Because there is also an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued.
21. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
22. Unresolved partial or complete small or large bowel obstruction
23. Judgment by the investigator that the patient is unsuitable to participate in the study or that the patient is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazaeri, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org